CLINICAL TRIAL: NCT07031479
Title: Efficacy of Enteral Itopride Versus Intravenous Metoclopramide in Hospitalized Medicine Patients With Feeding Intolerance Causing by High Gastric Residual Volume: a Prospective Randomized Controlled Trial
Brief Title: Efficacy of Itopride Versus Metoclopramide in Hospitalized Medicine Patients With High Gastric Residual Volume
Acronym: GRV
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0971/67
Record Dates: First submitted 2025-04-20; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-04

CONDITIONS: Feeding Intolerance
Keywords: gastric residual volume; metoclopramide; itopride
MeSH Terms: interventions — Metoclopramide

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Itopride (Experimental): Enteral Itopride (50 mg enterally tid ac)
  Interventions: Drug: Itopride HCI 50 mg
- Metoclopramide (Active Comparator): Intravenous Metoclopramide (10 mg IV q 6 hours)
  CrCl 15-60 ml/min: Metoclopramide 5 mg IV q 6 hours CrCl <15 ml/min: Metoclopramide 5 mg IV q 12 hours Hepatic impairment/ cirrhosis: Metoclopramide 5 mg IV q 6 hours
  Interventions: Drug: Metoclopramide 10 mg ampoule

INTERVENTIONS:
Drug: Itopride HCI 50 mg — Enteral Itopride 50 mg enterally tid ac
  Arms: Itopride
Drug: Metoclopramide 10 mg ampoule — Intravenous Metoclopramide (10 mg IV q 6 hours)
  CrCl 15-60 ml/min: Metoclopramide 5 mg IV q 6 hours CrCl <15 ml/min: Metoclopramide 5 mg IV q 12 hours Hepatic impairment/ cirrhosis: Metoclopramide 5 mg IV q 6 hours
  Arms: Metoclopramide

SUMMARY:
A prospective randomized controlled trial included 86 patients in medicine ward who were diagnosed with feeding intolerance, defined as having a gastric residual volume greater than 200 ml. The patients were randomly assigned to two treatment groups: one receiving enteral metoclopramide and the other receiving intravenous metoclopramide. The primary outcome was the gastric residual volume at 72 hours after treatment. The secondary outcome was gastric residual volume at 24 hours and 7 days after treatment, administered-to-prescribed volume at 72 hours after treatment, the administered-to-target energy ratio and the administered-to-target protein ratio at 96 hours after treatment, the nutrition status evaluated by the Nutrition Alert Form at 7 days after treatment, incidence of adverse events (arrhythmia, pneumonia, diarrhea, vomiting, aspiration), length of hospital stay, ICU length of stay and in-hospital mortality.

DETAILED DESCRIPTION:
Feeding intolerance was a significant problem commonly encountered during enteral feeding and led to cessation of enteral feeding. Prokinetics was recommended in feeding intolerance patients with a gastric residual volume greater than 200 ml, in conjunction with addressing underlying causes of gastrointestinal motility dysfunction, such as electrolyte imbalances and hyperglycemia. In Thailand, Metoclopramide was frequently used as the prokinetic of choice. However, its use was associated with significant adverse effects, including QTc interval prolongation and extrapyramidal symptoms. As a result, there was a limitation of Metoclopramide use in patients with a prolonged QTc interval. Itopride was a novel prokinetic agent which did not cause QTc prolongation and did not cross the blood-brain barrier. A randomized double-blind study conducted in ICU patients demonstrated that itopride significantly reduced GRV compared to the metoclopramide group. However, there was only one study focusing on ICU populations including both medicine and surgery patients. Therefore, the aim of our study was to evaluate the efficacy of itopride compared to metoclopramide in reducing gastric residual volume in medicine patients, including both ICU and non-ICU settings.

Our study was a prospective randomized controlled trial included 86 patients in medicine ward who were diagnosed with feeding intolerance, defined as having a gastric residual volume greater than 200 ml. The inclusion criteria were hospitalized medical patients aged over 18 years who were receiving enteral feeding and had a gastric residual volume (GRV) ≥ 200 ml. The exclusion criteria were use of any prokinetic drug within 24 hours before participating in the study, known hypersensitivity or contraindication to Metoclopramide or Itopride, prolonged QTc interval > 460 milliseconds in female or >440 milliseconds in male, hemodynamic instability, GI surgery ≤ 6 weeks before enrollment in the study, history of esophagectomy or gastrectomy, pregnancy, suspicious or confirmed gastrointestinal obstruction or gastrointestinal hemorrhage or gastrointestinal perforation, epilepsy or currently use of anti-epileptic drug, acute CNS infection or severe brain injury, Parkinson's disease, confirmed or suspected pheochromocytoma, history of tardive dyskinesia and history of methemoglobinemia.

The primary outcome of the study was the gastric residual volume at 72 hours after treatment. The secondary outcome was gastric residual volume at 24 hours and 7 days after treatment, administered-to-prescribed volume at 72 hours after treatment, the administered-to-target energy ratio and the administered-to-target protein ratio at 96 hours after treatment, the nutrition status evaluated by the Nutrition Alert Form at 7 days after treatment, incidence of adverse events (arrhythmia, pneumonia, diarrhea, vomiting, aspiration), length of hospital stay, ICU length of stay and in-hospital mortality.

The sample size was calculated to be 84 patients, using a minimum clinically important difference (MCID) of 50, a standard deviation of 77.6 (as referenced from a previous study), a 1:1 ratio, an alpha error of 5%, and a beta error of 20%.

After enrollment, all patients were evaluated for and treated for reversible causes of feeding intolerance, including electrolyte imbalances and hyperglycemia. Nutritional status was also assessed prior to the initiation of therapy. The patients were randomly assigned to two treatment groups: one receiving enteral metoclopramide and the other receiving intravenous metoclopramide. Patients received prokinetic therapy for 7 days. A stepwise advancement to full enteral feeding-targeted at 25-30 kcal/kg/day-was implemented by Day 4. The gastric residual volume was recorded four times daily, prior to feeding, and measured in milliliters. The gastric residual volume was measured manually by the nurse from a different team to maintain blinding in the administration of prokinetics. If the gastric residual volume (GRV) exceeded 200 ml for at least two instances per day, feeding advancement was withheld. The study termination criteria included an inability to advance feeding for 48 hours, a GRV ≥ 400 mL on two occasions, and a QTc interval > 440 ms in males and > 460 ms in females. Both the nurses and the doctors assessing the gastric residual volume (GRV) were blinded to the study conditions.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized medical patients aged over 18 years who were receiving enteral feeding and had a gastric residual volume (GRV) ≥ 200 ml

Exclusion Criteria:

* Use of any prokinetic drug within 24 hours before participating in the study
* Known hypersensitivity or contraindication to Metoclopramide or Itopride
* Prolonged QTc interval > 460 ms in female >440 ms in male
* Hemodynamic instability
* GI surgery ≤ 6 weeks before enrollment in the study
* History of esophagectomy or gastrectomy
* Pregnancy
* Suspicious or confirmed gastrointestinal obstruction or gastrointestinal hemorrhage or gastrointestinal perforation
* Epilepsy or currently use of anti-epileptic drug
* Acute CNS infection or severe brain injury
* Parkinson's disease
* Confirmed or suspected pheochromocytoma
* History of tardive dyskinesia, history of methemoglobinemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Mean gastric residual volume (in mL) on day 3 after initiation of prokinetics | Day3
  Mean gastric residual volume (in mL) on day 3 after initiation of prokinetics. The gastric residual volume was recorded four times daily, prior to feeding.

SECONDARY OUTCOMES:
Mean gastric residual volume (in mL) on day 1 after initiation of prokinetics | Day1
  Mean gastric residual volume (in mL) on day 1 after initiation of prokinetics. The gastric residual volume was recorded four times daily, prior to feeding.
Mean gastric residual volume (in mL) on day 7 after initiation of prokinetics | Day 7
  Mean gastric residual volume (in mL) on day 7 after initiation of prokinetics. The gastric residual volume was recorded four times daily, prior to feeding.
Percentage of prescribed enteral nutrition volume successfully administered on day 3 after initiation of prokinetics | Day 3
  Percentage of prescribed enteral nutrition volume successfully administered on day 3 after initiation of prokinetics.
  The goal total volume at day 3 was 1200 ml/day. (BD (1 kcal/1ml) 300 ml x 4 feed)
Percentage of target enteral nutrition energy successfully administered on day 4 after initiation of prokinetics | Day 4
  Percentage of target enteral nutrition energy (30 kcal/kg in non-ICU patients, 25 kcal/kg in ICU patients) successfully administered on day 4 after initiation of prokinetics
Percentage of target enteral nutrition protein successfully administered on day 4 after initiation of prokinetics | Day 4
  Percentage of target enteral nutrition protein (1.2 g/kg) successfully administered on day 4 after initiation of Prokinetics
Rate of participants experiencing adverse events (Percentage) | Up to 7 days
  Rate of participants experiencing adverse events (arrhythmia, pneumonia, diarrhea, vomiting, aspiration, abnormal movement)
Rate of In-Hospital mortality among Participants (Percentage) | Through study completion, an average of 1 year
  Rate of In-Hospital mortality among participants (Percentage), measured from the initiation of prokinetics to the time of discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Narisorn Lakananurak, MD., Study Director — Chulalongkorn University

IPD SHARING:
Plan to Share IPD: No